CLINICAL TRIAL: NCT04114682
Title: Longitudinal Assessment of Multiple Organs in Patients With Type 2 Diabetes
Acronym: MODIFY
Status: Active, not recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: University of Liverpool (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Oxford University Hospitals NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CA064
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; NAFLD; Metformin; Multiparametric MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Routine bloods will be performed as per standard-of-care for T2D; HbA1c, serum creatinine, electrolytes, lipids, FBC (full blood count), LFT (liver function tests (aspartate transaminase and alanine transaminase) and gamma glutamyl transferase (GGT) and eGFR.
  Additional circulating biomarkers, ie; the enhanced liver fibrosis test (ELF), N-terminal levels of type III procollagen (P3NP), pancreatic lipase, cystatin C, serum albumin, high sensitivity C-reactive protein, NT-proBNP and uric acid.
  Optional genetic testing for NAFLD or T2D associated genetic variants (serum sample).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multi parametric MRI scan — There will be no intervention to the standard of care these patients receive. However, consented participants will be asked to make two study visits where a multiparametric MRI scan will be performed - these visits will be defined as visit 2 and visit 3. An optional echocardiogram may be included at Visit 2.
  Other Names: Optional echocardiogram

SUMMARY:
MODIFY study is a multi-centre prospective, longitudinal, observational cohort study which aims to recruit 150 adult patients with type 2 diabetes recruited from community, primary care or secondary care settings. The total length of the study is 75 months. The aim of the study is to develop an MRI-based method to identify whom amongst people with Type 2 diabetes are at risk of further complications in their kidney, liver and cardiovascular system.

DETAILED DESCRIPTION:
There has been a surge in incidence of the metabolic syndrome; a cluster of conditions which increase the risk of, type 2 diabetes (T2D) (90% of diabetes cases), non-alcoholic fatty liver disease (NAFLD), non-alcoholic steatohepatitis (NASH), cardiovascular disease (including ischaemic heart disease and heart failure), ischaemic or haemorrhagic stroke

This project concentrates on T2D, a disease whose multiple patho-physiological defects include; increased renal glucose re-absorption, decreased peripheral glucose utilisation, increased hepatic glucose production due to insulin resistance, increased glucagon secretion, reduced insulin secretion (pancreas), and incretin secretion (gastrointestinal tract)

Estimated UK prevalence of T2D is 5.26%. This represents 3.3 million people (comparatively in the US, 9.1% or 26.44 million people), which equates to £8.8bn in associated healthcare costs in UK.

Type 2 diabetes is associated with a heterogeneity in its aetiology - this is observed in its clinical presentation and subsequent rate of progression. Further factors associated with T2D include micro-and macrovascular complications and an observed decline in multiple organs (end-organ damage). End-organ damage contributes to the clinical picture of individuals with T2D and is demonstrated when observing the high prevalence of co-morbidities in this patient cohort. For example, the presence of NAFLD is seen in 60% of T2D patients, along with a 34.2-50.7% presence of chronic kidney disease (CKD) and a 32.2% presence of cardiovascular disease (CVD).

Currently, T2D and its complications are monitored using circulating plasma and serum biomarkers. However, these lack sufficient sensitivity or specificity. An example of this is highlighted in one researcher's preliminary data that suggests that 85% of obese people with T2D had NAFLD, detected by MRI. However, a vast proportion of this patient cohort have recorded normal biochemical biomarkers, such as Alanine Transaminase (ALT).

Metformin is typically the initially treatment for T2D. However, due to its progressive nature, metformin monotherapy proves to be inadequate in maintaining long-term glycaemic control. Metformin has been used safely and effectively for decades, but newer drugs are becoming available. Numerous recent studies have shown that newer drug classes, including the SGLT-2 inhibitors and GLP1 receptor agonists (GLP-1RA), have substantial beneficial effects beyond modulation of glycaemic levels, and can confer protection against CVD and CKD. It is now recommended that use of these drugs is advocated for high risk populations with evidence of CKD or CVD.

This proposal aims to develop an MRI-based method that is able to identify the individuals at high risk of disease complications, looking particularly at renal, hepatic and cardiovascular pathology, and further compare this to the conventional biochemical approach. This has future potential in assisting in the stratification of patients to the most appropriate tailored treatment for their disease. The investigators will further evaluate the additional synergistic value of incorporating MRI-metrics into patient pathways.

There is a healthcare need to provide further decision-making support for clinicians in the care of patients at risk or diagnosed with T2D. This would combine multi-modality approaches, an incorporation of biochemical evaluation and imaging techniques. There is also a pressing need for treatment stratification to identify the T2D patients who would benefit from being triaged to receive the newer, more expensive drugs. This would also empower patients and aid in their engagement of the lifestyle changes often required for treatment. This should have the added benefit of reducing associated NHS costs by minimising the pool of patients with severe disease, who would be highlighted through early detection and early medical management.

To address this growing need, the investigators propose adding a complementary imaging aspect to the currently used biomarkers. MRI, specifically, provides excellent soft-tissue contrast. Perspectum's LiverMultiScan is a quantitative multiparametric MRI method, FDA-cleared and CE-marked, that is used to detect and stage early liver disease. It is already widely used in pharmaceutical trials for NAFLD therapeutics. The MRI metrics from LiverMultiScan can quantify changes to liver tissue characteristics, like fibro-inflammation and fat, as a result of intervention (for example, bariatric surgery). The accuracy and reproducibility of LiverMultiScan has been demonstrated in studies scanning patients within different MRI scanners. It continues to be further supported by data from clinical trials in liver disease cohorts, from comparative studies that include healthy controls, as well as whole-population studies in the UK and US.

With this proposal the investigators aim to develop a new MRI image analysis technique, "ATLAS", that builds on LiverMultiScan technology. the investigators also plan to gather clinical evidence that will demonstrate the potential added value to the NHS, as well as support future regulatory clearance. The phenotypical information that ATLAS delivers, combined with information from circulating biomarkers, will form the basis of a future clinical decision support tool for T2D.

Perspectum has pilot data showing that LiverMultiScan can estimate portal hypertension (spleen), detect pancreatitis, and characterise the tissue of the kidneys.

This proposal will extend LiverMultiScan to each of the other relevant organs - pancreas, kidneys and spleen. The technical development of "ATLAS" will be complemented by the accumulation and analysis of clinical data, circulating biomarkers and imaging. This information will be obtained from three diverse UK clinical centres (Liverpool, Oxford and London).

The innovation comes from combining a number of quantitative MRI metrics to achieve this:

* volumes - for liver, spleen, kidneys, pancreas;
* fibroinflammation: cT1 and/or T1 - for liver, spleen, kidneys, pancreas;
* fat infiltration: PDFF - for liver, kidneys, pancreas;
* aortic distensibility and diameter. The investigators will also incorporate kidney diffusion and renal flow. There will be strong patient and clinician involvement in the collection of patient-reported experience and outcome measures throughout the study (PREMs and PROMs), both qualitative and quantitative, to reflect the patients' experience of the clinical care pathway.

The resulting MRI diagnostic solution will enable rapid and comprehensive stratification of T2D and affiliated diseases (NAFLD, CKD, CVD), allowing clinicians to facilitate personalised medicine. It is anticipated that adopting a clinical approach which utilises ATLAS will result in substantial cost savings for the NHS and will help improve patient experience by providing access to advanced treatments to those patients most at risk.

The main objective of this study is to assess the health of multiple organs over a period of 9 months, using multiparametric abdominal MRI, in patients with type 2 diabetes who have been prescribed glucose lowering therapy (as per their standard of care).

This will be a multi-site study adopting a prospective, observational, longitudinal, cohort study design. There will be no intervention to the standard of care. Participants will be required to attend a screening visit and additional study visits on up to three time points - baseline (visit 1), a visit within 21 days of baseline (visit 2) and at 9-months (visit 3). The second and third visit will involve having a multiparametric MRI scan. Where possible, some visits (the screening visit visit 1 or visit 1 /visit 2) may be on the same day or within standard of care, depending on patient and MRI scanner availability.

Patients with type 2 diabetes and prescribed with glucose lowering therapy (as per standard of care) will be recruited from community settings, primary care centres and diabetes clinics within secondary care settings. The investigators aim to recruit patients who have been newly prescribed medication; also those patients undergoing treatment intensification (when an additional treatment is being considered due to evidence of poor glycaemic control), as per their standard of care HbA1c level results. Clinical outcome measurements, blood samples and urine samples will be collected to assess the response to standard of care treatment. There will be an optional thoracic echocardiogram (ECHO) included at visit 2. This is a non-invasive way in which the investigators can capture data to enable us to assess cardiovascular disease.

Study participants will be enrolled in this study for a total of 5-years. During this time, consented participants will be asked to attend for up to 3 study visits: Visit 1 (baseline), Visit 2 and Visit 3. Further to this, participants will be asked to give consent to the review of their medical records at 3 time points - years 1, 3, and 5, following baseline assessment. This review will be conducted by authorised study investigators who will obtain clinical outcome measures relating to the study objectives, for example, measures of liver or kidney function.

The primary endpoint of the study is to compare the MRI metrics for liver fibroinflammation in those patients with type 2 diabetes at baseline vs. individuals who are healthy and non-diabetic. Values for the healthy, non-diabetics will be provided from data from the UK Biobank (UKBB) and will be selected based on the matching of gender, age, ethnicity to the patients from this study with type 2 diabetes. Analysis will be based on a two-sample, two-sided t-test. The sample size required to perform a t-test with 90% power and alpha of 0.05 would require n=150.

Participants will be identified from the community, primary care and secondary care diabetes;appointments; specifically those patients with type 2 diabetes who are prescribed glucose lowering treatment as per their standard of care. A member of the clinical care team will provide potential participants with a study invitation letter and an accompanying Participant Information Leaflet (PIL) in the following places: Liverpool Diabetes Partnership/University Hospital Aintree, The Oxford Centre for Diabetes, Endocrinology and Metabolism (OCDEM) Oxford University Hospitals NHS Foundation Trust, The Royal Free London NHS Foundation Trust - Diabetes Department.

At each study centre, posters will be displayed around the hospitals, University departmental buildings and GP practices so that potential participants can also self-refer into the study by contacting the study team directly. The study will also be advertised on social media platforms (for example, Twitter and Facebook), Perspectum Diagnostics Ltd's website and also hospital websites. . Once a potential participant has been identified by any of these means, and has expressed an interest in taking part in the study, they will be sent a Participant Information Leaflet (PIL) to read. They will be allowed as much time as they require to understand the details of the study and what's involved before signing the consent form.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years of age and diagnosed with type 2 diabetes.
* Participant currently taking glucose lowering therapy.
* Participant willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (standard MR exclusion criteria including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Patients with known autoimmune hepatitis, viral hepatitis, Wilson's disease, haemoglobinopathies or significant structural renal tract abnormality.
* Patients with known excessive alcohol intake.
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants, aged 18 years and over, with type 2 diabetes and prescribed with glucose lowering therapy as per their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging metrics for liver fibro-inflammation in patients with type 2 diabetes | 1 year
  In order to determine the degree of liver fibro-inflammation in this cohort of patients with type 2 diabetes multi-parametric abdominal MRI will be performed. the measurements following the Multi parametric MRI in the type 2 diabetic patients will be compared with the same type of measurements in healthy individuals

SECONDARY OUTCOMES:
Correlation between Magnetic Resonance Imaging metrics for liver Fat infiltration and volume in patients with type 2 diabetes vs healthy people. | 1 year
  In order to determine the degree of liver fat infiltration and liver volume in this cohort of patients with type 2 diabetes, multi-parametric abdominal MRI will be performed. the measurements following the Multi parametric MRI in the type 2 diabetic patients will be compared with the same type of measurements in healthy individuals. in this way it could be also determine the proportion of people in this cohort with non-alcoholic fatty liver disease.
Correlation between Magnetic Resonance Imaging metrics for Pancreas, spleen, kidney and aorta indicating co-morbidities in patients with type 2 diabetes vs healthy people. | 1 year
  In order to determine the degree of abnormalities in other abdominal organs and aorta, in this cohort of patients with type 2 diabetes, multi-parametric abdominal MRI will be performed. The measurements following the Multi parametric MRI in the type 2 diabetic patients will be compared with the same type of measurements in healthy individuals. in this way it could be also determine the proportion of people in this cohort with non-alcoholic fatty liver disease.
Detecting change in liver, spleen, pancreas and kidney using Magnetic Resonance Imaging metrics from baseline to 9 months | 9 months
  To assess if multi-parametric abdominal MRI can quantify change in abdominal organs that occur over 9 months.
Detecting change in liver, spleen, pancreas and kidney using conventional biochemical biomarkers from baseline to 9 months | 9 months
  To assess changes in abdominal organs that occur over 9 months, with conventional biochemical biomarkers (glycaemic control, lipid profile, Creatinine, FBC and liver function tests) used in clinical pathway for patients with type 2 diabetes, chronic kidney disease and non alcoholic fatty liver disease.
Impact of Multi parametric abdominal MRI on management of patients with type 2 diabetes | 1 year
  To evaluate the effect multi parametric MRI has on the management of patients with type 2 diabetes, by reviewing and analysing patients and clinician reported outcome measures, using questionnaire
longer term evaluation of clinical outcomes | 5 years
  To determine the prognostic information provided by abdominal imaging for longer-term evaluation of clinical outcomes at 1 year, 3 years and 5 years. this includes assessing the odds ratio for developing cardiovascular, liver, pancreatic and kidney related events and / or death, including hospital admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cuthbertson, Study Chair — Liverpool hospitals
Locations (4):
- United Kingdom (4):
  - Aintree University Hospital NHS Foundation Trust, Liverpool, Merseyside
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Perspectum Ltd., Oxford, Oxfordshire
  - Royal Free Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT04114682/Prot_000.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04114682/ICF_001.pdf